CLINICAL TRIAL: NCT04481802
Title: The Effect of RadiaAce Gel Versus Biafine in the Prevention and Treatment of Radiation Dermatitis in Breast Cancer Patients
Brief Title: The Effect of RadiaAce Gel in the Prevention and Treatment of Radiation Dermatitis in Breast Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: AceTech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RadiaAce001
Record Dates: First submitted 2020-06-07; First posted 2020-07-22 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Breast Cancer; Radiation Dermatitis
Keywords: Radiation dermatitis; breast cancer
MeSH Terms: conditions — Breast Neoplasms; Radiodermatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RadiaAce gel (Experimental): RadiaAce Gel is a clear, non-oily Hydrogel wound dressing for the management of Radiation Dermatitis which provides optimal moist wound environment necessary to the healing process. RadiaAce gel contains Acemannan, a high molecular polysaccharide obtained from the inner gel of Aloe Vera leaves and it is considered the main functional component of Aloe vera (Sahu et al. 2013).
  Interventions: Device: RadiaAce gel
- Biafine (Active Comparator): one of the standard skin care in radiation oncology, this treatment was chosen as the comparator.
  Interventions: Device: Biafine

INTERVENTIONS:
Device: RadiaAce gel — Patients will apply the RadiaAce to the treatment area starting 5 days before radiation treatment. The Hydrogel/cream will be applied three times a day with a minimum of four hours between applications. Treatments will be used through the course of RT and for 6 days after the last fraction of radiation.
  Other Names: Acemannan hydrogel
  Arms: RadiaAce gel
Device: Biafine — Patients will apply the Biafine to the treatment area starting 5 days before radiation treatment. The Hydrogel/cream will be applied three times a day with a minimum of four hours between applications. Treatments will be used through the course of RT and for 6 days after the last fraction of radiation.
  Arms: Biafine

SUMMARY:
Radiation dermatitis (RD) is one of the most common side effects of Radiation therapy (RT) and 95% of patients receiving RT may experience some form of radiation dermatitis.

A wide variety of topical, oral, and intravenous agents are used to prevent/treat Radiation dermatitis but currently there is no gold standard in the prevention and management of this condition and no treatment can be explicitly recommended.

RadiaAce Gel is a wound dressing Hydrogel (Acemannan Hydrogel) for the management of RD which provides optimal moist wound environment necessary to the healing process.

Based on its composition as well as the supporting data on safety and performance of the functional ingredient Acemannan in wound healing, RadiaAce may well be suited to complement the prevention and therapy of radiation dermatitis.

The primary aim of the study is to evaluate the safety and performance of RadiaAce as compare to Biafine in reducing the proportion of breast cancer patients that experience grade 2 or higher RD as measured by the RTOG scoring system

ELIGIBILITY:
Inclusion Criteria:

1. Female patients
2. Age > 18
3. Patients with histologically-confirmed diagnosis of breast cancer
4. Patients after breast lumpectomy and that scheduled to receive radiotherapy
5. Patients to receive minimum of 40.05 Gy to primary field
6. Must be able to comply with treatment schedule
7. Study-specific signed informed consent prior to randomization

Exclusion Criteria:

1. Inflammatory or connective tissue disorders of the skin
2. Mental incompetence, including psychological or addictive disorders which would preclude completion of questionnaires
3. Previous radiation therapy to the breast
4. Tumour involvement of the skin
5. Rash, ulceration or open wound in treatment field
6. Known skin allergy or sensitivity to Aloe Vera or Biafine
7. Current lactation
8. Pregnancy
9. Any other reason that, in the opinion of the investigator, prevents the subject from

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-07-14 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Skin assessment (RD grade) | 10 weeks
  Skin condition (grade of RD) in the radiation area will be measured by the Radiation Therapy Oncology Group (RTOG) scoring
Pain (VAS) | 10 weeks
  Dermatitis-related pain is assessed with a visual analogue scale (VAS) self-assessment
Patient's assessment of the skin condition (DLQI questioner) | 10 weeks
  The Patients perspective is captured by the Dermatology Life Quality Index (DLQI)

CONTACTS AND LOCATIONS:
Overall Officials: Meirav Ben David, MD, Principal Investigator — Director of radiotherapy Institute
Locations (1):
- Assuta, Tel Aviv, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No